CLINICAL TRIAL: NCT00005898
Title: Phase I/II Study of Total Body Irradiation, Cyclophosphamide, and Fludarabine Followed by Alternate Donor Hematopoietic Cell Transplantation in Patients With Fanconi's Anemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/15109; UMN-MT-1999-05; UMN-MT9905
Record Dates: First submitted 2000-06-02; First posted 2000-06-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-07

CONDITIONS: Fanconi's Anemia
MeSH Terms: conditions — Fanconi Anemia | interventions — Antilymphocyte Serum; Cyclophosphamide; Cyclosporine; Filgrastim; fludarabine; Methylprednisolone

INTERVENTIONS:
Drug: anti-thymocyte globulin
Drug: cyclophosphamide
Drug: cyclosporine
Drug: filgrastim
Drug: fludarabine
Drug: methylprednisolone

SUMMARY:
OBJECTIVES: I. Determine the probability of engraftment with total body irradiation, cyclophosphamide, fludarabine, and anti-thymocyte globulin followed by HLA nongenotypically identical donor, T-cell depleted hematopoietic cell transplantation in patients with Fanconi's anemia.

II. Determine the incidence of acute and chronic graft-versus-host disease in these patients after undergoing this treatment regimen.

III. Determine the one-year survival rate in these patients after undergoing this treatment regimen.

IV. Determine the toxicity of this treatment regimen in these patients. V. Determine the incidence of relapse in patients with myelodysplastic syndrome or acute myeloid leukemia after undergoing this treatment regimen.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Donor bone marrow, peripheral blood, or umbilical cord blood is processed to harvest CD34+ cells.

Patients receive preparative cytoreductive therapy comprising total body irradiation on day -6; cyclophosphamide IV over 2 hours on days -5 to -2; fludarabine IV over 30 minutes on days -5 to -2; methylprednisone IV on days -5 to 24; anti-thymocyte globulin IV over 4-6 hours on days -5 to -1; cyclosporine IV over 2 hours every 12 hours (every 8 hours for patients less than 40 kg in weight) on days -3 to 180, and then tapering in the absence of graft-versus-host disease; hematopoietic cell transplantation on day 0; and filgrastim (G-CSF) IV starting on day 1 and continuing until blood counts recover.

Patients are followed at days 60, 90, and 180, and then annually for 3 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Patients with a diagnosis of Fanconi's anemia AND Aplastic anemia OR Myelodysplastic syndrome OR Acute leukemia with or without chromosomal anomalies Aplastic anemia as defined by having at least one of the following: Platelet count less than 20,000/mm3 Absolute neutrophil count less than 500/mm3 Hemoglobin less than 8 g/dL
* Myelodysplastic syndrome with multilineage dysplasia With or without chromosomal anomalies
* Hematologic malignancy (e.g., acute myeloid leukemia, acute lymphoblastic leukemia, or B-cell non-Hodgkin's lymphoma)
* No greater than 30% blasts in bone marrow or greater than 5% blasts in peripheral blood
* No active CNS leukemia at time of transplantation
* Must have an HLA A, B, DRB1 identical or 1 antigen mismatched related (nonsibling) or unrelated bone marrow, peripheral blood, or umbilical cord blood donor

--Prior/Concurrent Therapy--

* Radiotherapy: No prior radiotherapy that would preclude total body irradiation
* Surgery: Not specified

--Patient Characteristics--

* Performance status: Karnofsky 70-100% OR Lansky 50-100%
* Hematopoietic: See Disease Characteristics
* Hepatic: No hepatic failure (e.g., coagulopathy or ascites)
* Renal: Creatinine clearance at least 40 mL/min
* Cardiovascular: Ejection fraction at least 45%
* Other: No active uncontrolled infection within one week of transplantation No malignant solid tumor (e.g., squamous cell carcinoma of the head, neck, or cervix) within 2 years of transplantation Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

Ages: 0 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30
Dates: Start 2000-02

CONTACTS AND LOCATIONS:
Overall Officials: John E. Wagner, Jr., Study Chair — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Cancer Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] MacMillan ML, DeFor TE, Young JA, Dusenbery KE, Blazar BR, Slungaard A, Zierhut H, Weisdorf DJ, Wagner JE. Alternative donor hematopoietic cell transplantation for Fanconi anemia. Blood. 2015 Jun 11;125(24):3798-804. doi: 10.1182/blood-2015-02-626002. Epub 2015 Mar 30. PMID 25824692